CLINICAL TRIAL: NCT00107562
Title: Adolescent Safer Sex Social Network Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATN 032
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: Sexual Behavior; Alcohol Drinking; Marijuana Smoking
Keywords: risk behavior; social networks; behavior
MeSH Terms: conditions — Sexual Behavior; Alcohol Drinking; Marijuana Smoking; Risk-Taking; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): The cohort will be comprised of up to 4 index participants and from 1-4 of their network members for a possible range of 8-16 subjects in each cohort (average of 12 per cohort). The vast majority of the intervention will be delivered to both females and males together, but it would be beneficial, and appropriate for this adolescent population, to deliver certain exercises with the two genders separated.
  Interventions: Behavioral: Adolescent Safer Sex Social Network Intervention

INTERVENTIONS:
Behavioral: Adolescent Safer Sex Social Network Intervention

SUMMARY:
Social networks are thought to hold the potential for shaping behavior on the grounds that social and situational factors more strongly influence behavior than do personality variables. This is a behavioral intervention study that will test a 6-session, small-group, peer-network intervention among adolescent males and females and their friends. The intervention primarily focuses on reducing risky sexual behavior and increasing condom use among adolescent males and females, aged 16-19. The concurrent use of alcohol and marijuana during sex is also a focus as these two substances are widely used among adolescents and fuel risky sexual behavior.

DETAILED DESCRIPTION:
The objective of this Phase II study is to test the feasibility, acceptability and preliminary effectiveness of a 6-session, small-group, peer-network intervention among adolescent males and females and their friendship networks.

A one-arm intervention design with pre-test assessment within one month before the first intervention session, and with post-test assessments at three and six months following intervention completion will be used. The intervention will be delivered to cohorts of friendship groups comprised of an index friend and their social network. To ensure that baseline data reflect recent, pre-intervention behavior, index participants and their networks will be recruited in small 'cohorts' of 8-16 (average 12) adolescents at a time. These cohorts will then receive the group intervention at the same time. Each cohort of interested and eligible participants (index + network members) will be screened and consented, and will provide baseline data. The first intervention session must occur within one month of baseline data collection. A successive series of these small cohorts will be identified, enrolled and dispatched to receive the intervention with subsequent follow up timelines determined by the date of the final group session of each cohort.

Preliminary effectiveness of the behavioral intervention will be measured as follows:

* The primary outcome related to sexual behavior is the self-reported number of unprotected (not protected with male or female condom) vaginal, oral and anal sex acts among all (index and network members) who receive the intervention.
* Sexual acts when drunk or high will be measured by counting the number of sexual encounters that occurred concurrently with a respondent reporting being "drunk" or "high".
* Alcohol use will be measured by calculating the mean number of drinks consumed. Data will be collected on:

  * the overall frequency of alcohol consumption during the referent period (past 3 months); and
  * the usual number of drinks consumed on days when the individual reported drinking alcohol.

The network effect on sexual and drug-use behaviors will be measured as follows:

* Data at each of the three time points (baseline, 3 and 6 months) will be evaluated to determine whether sexual and drug-use behaviors within networks are more correlated than such behaviors between networks.

ELIGIBILITY:
Inclusion Criteria:

Index Participant Inclusion Criteria

* Self-identifies as all or part "Latino"
* Age is between 16 years and 0 days and 19 years and 364 days at the time of study enrollment
* In the past 3 months, reports engaging in any type of heterosexual sex (vaginal, oral or anal) with an opposite-sex partner
* In the past 3 months, reports any of the following:

  * alcohol use at least once;
  * marijuana use at least once;
  * having sex while drunk or high.
* Must understand spoken and written English sufficiently to provide consent/assent and be interviewed and attend intervention workshops delivered in English
* Must live in the Boston or Tampa area, and plan to be available for study appointments (vacation allowed if not interfering with the planned intervention or follow up dates)

Network Participant Inclusion Criteria

* Age is between 16 years and 0 days to 19 years and 364 days at the time of study enrollment
* In the past 3 months, reports engaging in any type of heterosexual sex (vaginal, oral or anal) with an opposite-sex partner
* Must understand spoken and written English sufficiently to provide consent/assent and be interviewed and attend intervention workshops delivered in English
* Must live in the Boston or Tampa area, and plan to be available for study appointments (vacation allowed if not interfering with the planned intervention or follow up dates)
* Must be reported by an index as a friend who:

  * has been known for at least 6 months;
  * hangs out with, or is in contact with the index at least 2 times per week;
  * has engaged in alcohol or marijuana use with the index during the last 3 months; and
  * gave directive guidance (gave index information on how to do something) AND, had intimate interaction (i.e. listened to private feelings of index) AND, had positive social interaction with the index.

Exclusion Criteria:

Index Participant Exclusion Criteria

* Reports only same sex behavior
* Reports being HIV positive, as measured by self-report
* Reports having engaged in behaviors in the past year that are defined as "severe" physical abuse of others on the Conflict Tactics Scale
* In the past year, reports having made someone engage in sexual things that he or she did not want to do either by holding the partner down, hurting or by threatening them in some way
* Unable to nominate at least one eligible friend to participate in the intervention
* Reports having ever used heroin, crack, cocaine, or metamphetamines
* Reports alcohol dependence as measured by affirmative answers to 3 or more out of 7 questions on the Diagnostic and Statistical Manual of Mental Disorders - 4th Edition (DSM-IV) based criteria of substance dependence
* Reports marijuana dependence as measured by affirmative answers to 3 or more out of 7 questions on the DSM-IV based criteria of substance dependence
* Reports being an active member of a gang
* Reports or is known by staff to be currently participating in any other bio-medical or Adolescent Trial Network (ATN)-related intervention study or trial
* If female, reports being currently pregnant
* Unwilling to be screened for sexually transmitted infections (STIs)
* Prior participation in this study intervention as either an index or a network member as determined by review of study logs

Network Participant Exclusion Criteria

* Is currently romantically involved with the index who named him/her
* Has ever had vaginal, oral or anal sex with the index
* Reports only same sex behavior
* Reports being HIV positive, as measured by self-report
* Reports having engaged in behaviors in the past year that are defined as "severe" physical abuse of others on the Conflict Tactics Scale
* In the past year, reports having made someone engage in sexual things that he or she did not want to do either by holding the partner down, hurting or by threatening him/her in some way
* Reports having ever used heroin, crack, cocaine, or metamphetamines
* Reports alcohol dependence as measured by affirmative answers to 3 or more out of 7 questions on the DSM-IV based criteria of substance dependence
* Reports marijuana dependence as measured by affirmative answers to 3 or more out of 7 questions on the DSM-IV based criteria of substance dependence
* Self-reports being an active member of a gang
* Reports or is known by staff to be currently participating in any other bio-medical or ATN-related intervention study or trial
* If female, reports being currently pregnant
* Unwilling to be screened for STIs
* Prior participation in this study intervention as either an index or a network participant as determined by review of study logs

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2005-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Test the feasibility, acceptability and preliminary effectiveness intervention | 6 Months
  The objective of this Phase II study is to test the feasibility, acceptability and preliminary effectiveness of a 6-session, small-group, peer-network intervention among adolescent males and females and their friendship networks. The ultimate goal is to test the intervention in a randomized, attention-controlled, Phase III trial.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Latka, PhD, Study Chair — New York Academy of Medicine
Locations (2):
- United States (2):
  - University of South Florida College of Medicine, Tampa, Florida
  - Children's Hospital of Boston, Boston, Massachusetts

REFERENCES:
- See also: description of the Adolescent Trials Network and contact information — http://www.atnonline.org